CLINICAL TRIAL: NCT00949871
Title: Sister Survivor: African American Breast Cancer Coalition
Brief Title: Study of Support Groups for African-American Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None
Other Study IDs: 07170; P30CA033572 (NIH); CHNMC-07170; CDR0000642441 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Cancer Survivor
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; cancer survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: communication analysis
Other: questionnaire administration
Procedure: psychosocial assessment and care
Procedure: support group therapy

SUMMARY:
RATIONALE: A study that evaluates successful Los Angeles-based, peer-led African American breast cancer survivor support groups may help in developing a guide on how to organize and maintain breast cancer support groups.

PURPOSE: This clinical trial is studying support groups for African-American breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterize five established Los Angeles (LA)-based, peer-led African American Breast Cancer Survivor (AABCS) support groups by identifying and evaluating the successful elements of structure and process that distinguish these groups: the purpose and goals; theories and techniques that are utilized; the structure of the group and implementation of specific goals; the cultural aspects that are incorporated to enhance the efficacy; and similarities and differences among these AABCS support groups.
* Develop a preliminary "Culturally Informed Breast Cancer Support Group Guide" on how to organize and maintain support groups, modeled on the "best model" experiences of the five established LA-based support groups for AABCS.
* Conduct three needs-assessment focus groups and 5 key informant interviews in the Inland Empire to evaluate the psychosocial needs and resources of AABCS in that region.

OUTLINE: At least 10 support group leaders (2 from each support group) undergo semi-structured interviews to elicit information about the needs of breast cancer survivors in their community and the cultural modes of support that are given. Eight to twelve African American Breast Cancer Survivors (AABCS) participate in 5 focus group discussions and complete a questionnaire about their breast cancer and experience with support groups for qualitative and quantitative analysis.

At least 5 Inland Empire community leaders undergo semi-structured interviews to elicit information about the needs of breast cancer survivors in their community. Eight to twelve AABCS from the Inland Empire participate in 3 focus group discussions and complete a questionnaire about their breast cancer and experience with support groups for qualitative and quantitative analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * African American Breast Cancer Survivor (AABCS) meeting 1 of the following criteria:

    * A member of 1 of the 5 support groups listed below
    * Live in the Inland Empire region of California
  * A cancer support group leader or facilitator of 1 of the 5 established support groups in Los Angeles:

    * Women of Essence (WOE)
    * Women of Color (WOC)
    * Support Sisters African American Breast Cancer Support Groups
    * Sisters
    * Celebrate Life
  * A community leader knowledgeable about breast cancer support services in the Inland Empire region

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Characterization of five established Los Angeles-based, peer-led African American Breast Cancer Survivor (AABCS) support groups
Preliminary "Culturally-Informed Breast Cancer Support Group Guide" on how to organize and maintain support groups
Completion of 3 needs-assessment focus group sessions and 5 key-informant interviews in the Inland Empire

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States